CLINICAL TRIAL: NCT07072637
Title: A Prospective Study Assessing Neurological Function and Its Clinical Implications in Patients With Locally Advanced or Metastatic Urothelial Carcinoma Receiving Enfortumab Vedotin-Based Therapy
Brief Title: Neurological Function in Patients With Locally Advanced or Metastatic Urothelial Carcinoma Treated With Enfortumab Vedotin-Based Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202502005RINB
Record Dates: First submitted 2025-06-29; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced or Metastatic Urothelial Carcinoma
Keywords: enfortumab vedotin; urothelial carcinoma; neurological function
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EV-based therapy: Patients with locally advanced or metastatic urothelial carcinoma receiving enfortumab vedotin-based therapy
  Interventions: Diagnostic Test: Neurological function assessment

INTERVENTIONS:
Diagnostic Test: Neurological function assessment — Neurological evaluations including neurological examination (NE), nerve conduction study (NCS), quantitative sensory testing (QST), autonomic function testing (AFT), and the Toronto Clinical Neuropathy Score (TCNS) questionnaire. Assessments will be conducted at baseline and every three months until six months after completion of EV treatment.

SUMMARY:
This prospective observational study aims to evaluate the correlation between neurological function and patient-reported symptoms of peripheral neuropathy (PN) in patients with locally advanced or metastatic urothelial carcinoma (la/mUC) receiving enfortumab vedotin (EV)-based therapy. A total of 100 patients will be enrolled between March 2025 and December 2029. Eligible participants will undergo comprehensive neurological assessments, including neurological examination(NE), nerve conduction study (NCS), quantitative sensory testing (QST), autonomic function testing (AFT), and the Toronto Clinical Neuropathy Score (TCNS) questionnaire. These assessments will be conducted at baseline and every three months until six months after completion of EV-based therapy. Patient characteristics and oncological outcomes will also be collected. This study seeks to identify risk factors for developing PN and to explore the clinical implications of EV-associated neurological changes, with the ultimate goal of optimizing treatment strategies and improving quality of life.

DETAILED DESCRIPTION:
Peripheral neuropathy (PN) is a frequent and often debilitating adverse event associated with enfortumab vedotin (EV), a NECTIN-4-directed antibody-drug conjugate approved for patients with locally advanced or metastatic urothelial carcinoma (la/mUC). While EV has demonstrated significant antitumor efficacy, the objective assessment of PN and its clinical implications remain insufficiently explored. This prospective observational study aims to comprehensively evaluate neurological function and its correlation with subjective PN symptoms in la/mUC patients receiving EV-based therapy.

A total of 100 patients will be prospectively enrolled between March 2025 and December 2029. Neurological assessments will include neurological neurological examination (NE), nerve conduction study (NCS), quantitative sensory testing (QST), autonomic function testing (AFT), and the Toronto Clinical Neuropathy Score (TCNS) questionnaire. These evaluations will be conducted at baseline and every three months until six months post-EV treatment. Clinical data, including patient characteristics and oncologic outcomes, will also be collected.

This study aims to identify predictive factors for EV-related PN and to evaluate the broader clinical implications of neurological function changes. The ultimate goal is to inform strategies for toxicity mitigation and to optimize therapeutic outcomes and quality of life in la/mUC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 y/o
2. Histologically confirmed urothelial carcinoma
3. Radiologically documented locally advanced or metastatic disease
4. Prepare for receiving EV (as monotherapy or in combination with immune checkpoint inhibitors)
5. Complete and identifiable medical records

Exclusion Criteria:

1. Do not agree to receive regular neurological examinations
2. Do not agree to provide complete medical records during treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥ 20 years) with histologically confirmed locally advanced or metastatic urothelial carcinoma who are planned to receive EV-based therapy. Participants must be eligible for neurological assessments and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between neurological function and subjective peripheral neuropathy symptoms | Baseline to 6 months post-treatment.
  Correlation between objective neurological assessments (nerve conduction study, QST, autonomic function tests, TCNS) and patient-reported peripheral neuropathy symptoms.

SECONDARY OUTCOMES:
Correlation between neurological function changes and oncological outcomes | From date of EV initiation to the date of death from any cause, assessed up to 36 months
  To evaluate whether the degree or pattern of neurological function changes (e.g., worsening in NCS, QST) correlates with clinical efficacy measures such as objective response rate (ORR), progression-free survival (PFS), and overall survival (OS).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT07072637/Prot_000.pdf